CLINICAL TRIAL: NCT02659059
Title: A Study of Nivolumab in Combination With Ipilimumab (Part 1); and Nivolumab Plus Ipilimumab in Combination With Chemotherapy (Part 2) as First Line Therapy in Stage IV Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Nivolumab in Combination With Ipilimumab (Part 1); Nivolumab Plus Ipilimumab in Combination With Chemotherapy (Part 2) as First Line Therapy in Stage IV Non-Small Cell Lung Cancer
Acronym: CheckMate 568
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-568
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Results first posted 2021-07-22 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Ipilimumab; CP protocol; Cisplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab+Ipilimumab (Experimental): Part 1
  Specified Dose on Specified Days
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Nivolumab+Ipilimumab + 2 cycles Platinum Doublet Chemotherapy (Experimental): Part 2
  Specified Dose on Specified Days
  Interventions: Biological: Nivolumab; Biological: Ipilimumab; Drug: Platinum Doublet Chemotherapy

INTERVENTIONS:
Biological: Nivolumab — Specified Dose on Specified Days
  Other Names: BMS-936558; Opdivo
Biological: Ipilimumab — Specified Dose on Specified Days
  Other Names: BMS-734016; Yervoy
Drug: Platinum Doublet Chemotherapy
  Other Names: Carboplatin + Paclitaxel; Cisplatin + pemetrexed
  Arms: Nivolumab+Ipilimumab + 2 cycles Platinum Doublet Chemotherapy

SUMMARY:
The purpose of part 1 of this study is to determine the objective response rate (ORR) in stage IV NSCLC subjects treated with nivolumab in combination with ipilimumab as first line therapy.

The purpose of part 2 of this study is to determine the safety and tolerability of nivolumab and ipilimumab combined with a short course of chemotherapy in first line stage IV NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women ≥ 18 years of age
* Diagnosed with stage IV Non-Small Cell Lung Cancer
* Diagnosed with recurrent stage IIIB non-small cell lung cancer and failed previous concurrent chemoradiation with no further curative options.

Exclusion Criteria:

* Subjects with untreated CNS metastases are excluded.
* Subjects with carcinomatous meningitis
* Subjects with an active, known or suspected autoimmune disease.
* Subjects with a condition requiring systemic treatment with either corticosteroids ( > 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first treatment.
* Women who are pregnant, plan to become pregnant, and/or breastfeed during the study.

Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2022-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (32):
- United States (29):
  - Sharp Memorial Hospital, San Diego, California
  - Cancer Center Of Central Connecticut, Plainville, Connecticut
  - Cleveland Clinic Florida, Weston, Florida
  - Winship Cancer Institute., Atlanta, Georgia
  - Summit Cancer Care, Savannah, Georgia
  - Cancer Center Of Kansas, Wichita, Kansas
  - University Of Louisville Medical Center, Inc., Dba, Louisville, Kentucky
  - Johns Hopkins Cancer Center, Baltimore, Maryland
  - Local Institution - 0029, Boston, Massachusetts
  - Local Institution - 0030, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Local Institution - 0015, Lincoln, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Local Institution - 0036, Albuquerque, New Mexico
  - Lovelace Cancer Care, Albuquerque, New Mexico
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - New Mexico Cancer Care Center, Albuquerque, New Mexico
  - The Cancer Center at Presbyterian, Albuquerque, New Mexico
  - Local Institution - 0010, Mineola, New York
  - Memorial Sloan Kettering Nassau, New York, New York
  - Duke University, Durham, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Local Institution - 0006, Pittsburgh, Pennsylvania
  - Charleston Hematology Oncology Associates, Pa, Charleston, South Carolina
  - Tennessee Oncology, PLLC - SCRI - PPDS, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Canada (3):
  - Local Institution - 0022, Kingston, Ontario
  - Local Institution - 0023, Sault Ste. Marie, Ontario
  - Csss De St-Jerome, Saint-Jérôme, Quebec

REFERENCES:
- [Derived] Ready N, Hellmann MD, Awad MM, Otterson GA, Gutierrez M, Gainor JF, Borghaei H, Jolivet J, Horn L, Mates M, Brahmer J, Rabinowitz I, Reddy PS, Chesney J, Orcutt J, Spigel DR, Reck M, O'Byrne KJ, Paz-Ares L, Hu W, Zerba K, Li X, Lestini B, Geese WJ, Szustakowski JD, Green G, Chang H, Ramalingam SS. First-Line Nivolumab Plus Ipilimumab in Advanced Non-Small-Cell Lung Cancer (CheckMate 568): Outcomes by Programmed Death Ligand 1 and Tumor Mutational Burden as Biomarkers. J Clin Oncol. 2019 Apr 20;37(12):992-1000. doi: 10.1200/JCO.18.01042. Epub 2019 Feb 20. PMID 30785829
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 324 participants treated
Groups:
- Nivolumab+Ipilimumab: Part 1 Nivolumab IV 3 mg/kg Q2W + Ipilimumab IV 1 mg/kg Q6W
- Nivolumab+Ipilimumab+Chemotherapy: Part 2 Nivolumab IV 360mg Q3W + Ipilimumab IV 1 mg/kg Q6W + 2 cycles Platinum Doublet Chemotherapy
Period: Overall Study
Arm/Group | Nivolumab+Ipilimumab | Nivolumab+Ipilimumab+Chemotherapy
Started | 288 | 36
Completed | 37 | 4
Not Completed | 251 | 32
Not completed — Other reasons | 6 | 1
Not completed — Disease Progression | 143 | 16
Not completed — Study Drug toxicity | 56 | 9
Not completed — Death | 3 | 1
Not completed — Adverse Event unrelated to Study drug | 32 | 4
Not completed — Participant request to discontinue study treatment | 5 | 0
Not completed — Participant withdrew consent | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab+Ipilimumab | Nivolumab+Ipilimumab+Chemotherapy | Total
Number analyzed (Participants) | 288 | 36 | 324
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 135 | 13 | 148
  >=65 years | 153 | 23 | 176
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 13 | 159
  Male | 142 | 23 | 165
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 0 | 12
  Not Hispanic or Latino | 258 | 36 | 294
  Unknown or Not Reported | 18 | 0 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 4 | 23
  White | 259 | 32 | 291
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) by PD-L1 Positive and Negative Levels - Part 1
Description: Objective response rate (ORR) in PD-L1 positive (PD-L1 ≥1%) and PD-L1 negative (PD-L1 <1%) participants was defined as the percentage of treated participants with confirmed complete response (CR) or partial response (PR) per RECIST 1.1 based on Blinded Independent Central Review (BICR) assessment.
Time Frame: From first dose to database lock (Up to 18 months)
Population: All PD-L1 evaluable participants -Part 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab+Ipilimumab
Number analyzed (Participants) | 252
Percentage of participants
  PD-L1 ≥1%: number analyzed (Participants) | 138
  PD-L1 ≥1% | 41.3 [33.0 to 50.0]
  PD-L1 <1%: number analyzed (Participants) | 114
  PD-L1 <1% | 14.9 [8.9 to 22.8]

2. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) - Part 2
Description: Dose limiting toxicities (DLTs) were defined as any of the items listed below.
  1. Any Grade 2 drug-related uveitis or eye pain that does not respond to topical therapy and does not improve to Grade 1 severity within the re-treatment period OR requires systemic treatment.
  2. Any Grade 2 drug-related pneumonitis or interstitial lung disease that does not resolve to dose delay and systemic steroids in 14 days.
  3. Any Grade 3 non-skin drug-related adverse event with the exception of laboratory abnormalities that cannot be alleviated or controlled by appropriate care within 14 days.
  4. Any Grade 4 drug-related adverse event including laboratory abnormalities except Grade 4 leukopenia or neutropenia lasting < 14 days and asymptomatic amylase/lipase elevation.
  5. Drug-related hepatic function laboratory abnormalities.
Time Frame: 9 weeks after first dose
Population: All treated participants -Part 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab+Ipilimumab+Chemotherapy
Number analyzed (Participants) | 36
Participants | 1

3. Primary Outcome: Number of Participants With Adverse Events (AEs) - Part 2
Description: Number of participants with adverse events (AEs) including serious adverse events (SAEs) and deaths graded by Common Terminology Criteria for Adverse Events (CTCAE v4.0) to determine the safety and tolerability of Nivolumab and Ipilimumab combined with chemotherapy.
Time Frame: Deaths are from first dose to database lock (Up to 24 months). AEs and SAEs are from first dose to 30 days post last dose
Population: All treated participants -Part 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab+Ipilimumab+Chemotherapy
Number analyzed (Participants) | 36
Participants
  Adverse Events (AEs) | 36
  Serious Adverse Events (SAEs) | 26
  Deaths due to Disease progression | 9
  Deaths due to Study drug toxicity | 0
  Deaths due to unknown causes | 1
  Deaths due to other causes | 6

4. Primary Outcome: Number of Participants With Laboratory Abnormalities in Hepatic Tests - Part 2
Description: Number of participant with specific liver laboratory abnormalities graded by Common Terminology Criteria for Adverse Events (CTCAE v4.0) to determine the safety and tolerability of Nivolumab and Ipilimumab combined with chemotherapy.
Time Frame: From first dose to 30 days post last dose
Population: All treated participants with at least one on-treatment measurement of the corresponding laboratory parameter -Part 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab+Ipilimumab+Chemotherapy
Number analyzed (Participants) | 35
Participants
  ALT OR AST >3XULN | 2
  ALT OR AST >5XULN | 2
  ALT OR AST >10XULN | 1
  ALT OR AST >20XULN | 1
  TOTAL BILIRUBIN >2XULN | 0
  Concurrent ALT OR AST >3XULN & BILIRUBIN >2XULN within 1 day | 0
  Concurrent ALT OR AST >3XULN & BILIRUBIN >2XULN within 30 days | 0

5. Primary Outcome: Number of Participants With Laboratory Abnormalities in Thyroid Tests - Part 2
Description: Number of participants with specific thyroid laboratory abnormalities graded by Common Terminology Criteria for Adverse Events (CTCAE v4.0) to determine the safety and tolerability of Nivolumab and Ipilimumab combined with chemotherapy.
Time Frame: From first dose to 30 days post last dose
Population: All treated participants with at least one on-treatment TSH measurement -Part 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab+Ipilimumab+Chemotherapy
Number analyzed (Participants) | 34
Participants
  TSH > ULN | 10
  TSH > ULN with TSH <= ULN at baseline | 7
  TSH > ULN with at least one FT3/FT4 test value < LLN | 8
  TSH > ULN with all other FT3/FT4 test values ≥ LLN | 1
  TSH > ULN with FT3/FT4 test missing | 1
  TSH < LLN | 13
  TSH < LLN with TSH >= LLN at baseline | 12
  TSH < LLN with at least one FT3/FT4 test value > ULN | 7
  TSH < LLN with all other FT3/FT4 test values <= ULN | 6
  TSH < LLN with FT3/Ft4 test missing | 0

6. Secondary Outcome: Overall Survival (OS) - Part 1
Description: Overall survival (OS) was defined as the time from date of first treatment to the date of death due to any cause. A participant who has not died will be censored at the last known date alive.
Time Frame: From the date of first treatment to the date of death due to any cause (Up to approximately 72 months)
Population: All treated participants in Part 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab+Ipilimumab
Number analyzed (Participants) | 288
Months | 20.83 [14.46 to 25.20]

7. Secondary Outcome: Overall Survival (OS) - Part 2
Description: as for outcome 6
Time Frame: From the date of first treatment to the date of death due to any cause (Up to approximately 59 months)
Population: All treated participants in Part 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab+Ipilimumab+Chemotherapy
Number analyzed (Participants) | 36
Months | 19.35 [6.54 to 35.42]

8. Secondary Outcome: Progression Free Survival (PFS) - Part 1
Description: Progression Free Survival (PFS) was defined as the time between the date of first dose and the first date of documented progression, as determined by blinded independent central review (BICR), or death due to any cause, whichever occurred first. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From first dose to the first date of documented progression, or death due to any cause, whichever occurred first (Up to approximately 72 months)
Population: All treated participants in Part 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab+Ipilimumab
Number analyzed (Participants) | 288
Months | 5.19 [3.06 to 5.82]

9. Secondary Outcome: Progression Free Survival (PFS) - Part 2
Description: Progression Free Survival (PFS) was defined as the time between the date of first dose and the first date of documented progression, as determined by investigator (per RECIST 1.1), or death due to any cause, whichever occurred first. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From first dose to the first date of documented progression, or death due to any cause, whichever occurred first (Up to approximately 59 months)
Population: All treated participants in Part 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab+Ipilimumab+Chemotherapy
Number analyzed (Participants) | 36
Months | 10.81 [5.26 to 16.13]

10. Secondary Outcome: Objective Response Rate (ORR) - Part 1
Description: Objective response rate (ORR) was defined as the percentage of treated participants with confirmed complete response (CR) or partial response (PR) per RECIST 1.1 based on Blinded Independent Central Review (BICR) assessment.
  CR = Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  PR = At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose up to approximately 72 months
Population: All treated participants in Part 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab+Ipilimumab
Number analyzed (Participants) | 288
Percentage of participants | 32.3 [26.9 to 38.0]

11. Secondary Outcome: Objective Response Rate (ORR) - Part 2
Description: Objective response rate (ORR) was defined as the percentage of treated participants with confirmed complete response (CR) or partial response (PR) per RECIST 1.1 based on investigator assessment.
  CR = Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  PR = At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose up to approximately 59 months
Population: All treated participants in Part 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab+Ipilimumab+Chemotherapy
Number analyzed (Participants) | 36
Percentage of participants | 47.2 [30.4 to 64.5]

12. Secondary Outcome: Overall Survival (OS) by PD-L1 Expression Levels - Part 1
Description: Overall survival (OS) by PD-L1 expression levels was defined as the time from date of first treatment to the date of death due to any cause. A participant who has not died will be censored at the last known date alive.
  PD-L1 ≥1% = PD-L1 positive (membranous staining in ≥ 1% tumor cells) PD-L1 <1% = PD-L1 negative (membranous staining in <1% tumor cells)
Time Frame: From the date of first treatment to the date of death due to any cause (Up to approximately 72 months)
Population: All PD-L1 evaluable participants in Part 1. Data was pre-specified to be collected only in Part 1 arm
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab+Ipilimumab
Number analyzed (Participants) | 255
Months
  PD-L1 ≥1%: number analyzed (Participants) | 138
  PD-L1 ≥1% | 26.51 [17.12 to 43.17]
  PD-L1 <1%: number analyzed (Participants) | 117
  PD-L1 <1% | 13.70 [10.71 to 21.91]

13. Secondary Outcome: Progression Free Survival (PFS) by PD-L1 Expression Levels - Part 1
Description: Progression Free Survival (PFS) by PD-L1 expression levels was defined as the time between the date of first dose and the first date of documented progression, as determined by blinded independent central review (BICR), or death due to any cause, whichever occurred first. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  PD-L1 ≥1% = PD-L1 positive (membranous staining in ≥ 1% tumor cells) PD-L1 <1% = PD-L1 negative (membranous staining in <1% tumor cells)
Time Frame: as for outcome 8
Population: All PD-L1 evaluable participants in Part 1. Data was pre-specified to be collected only in Part 1 arm
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab+Ipilimumab
Number analyzed (Participants) | 255
Months
  PD-L1 ≥1%: number analyzed (Participants) | 138
  PD-L1 ≥1% | 6.80 [4.17 to 10.97]
  PD-L1 <1%: number analyzed (Participants) | 117
  PD-L1 <1% | 2.92 [2.17 to 4.11]

14. Secondary Outcome: Objective Response Rate (ORR) by PD-L1 Expression Levels-Part 1
Description: Objective response rate (ORR) by PD-L1 expression levels was defined as the percentage of treated participants with confirmed complete response (CR) or partial response (PR) per RECIST 1.1 based on Blinded Independent Central Review (BICR) assessment.
  CR = Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  PR = At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  PD-L1 ≥1% = PD-L1 positive (membranous staining in ≥ 1% tumor cells) PD-L1 <1% = PD-L1 negative (membranous staining in <1% tumor cells)
Time Frame: From first dose up to approximately 72 months
Population: All PD-L1 evaluable participants in Part 1. Data was pre-specified to be collected only in Part 1 arm
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab+Ipilimumab
Number analyzed (Participants) | 255
Percentage of participants
  PD-L1 ≥1%: number analyzed (Participants) | 138
  PD-L1 ≥1% | 44.2 [35.8 to 52.9]
  PD-L1 <1%: number analyzed (Participants) | 117
  PD-L1 <1% | 17.1 [10.8 to 25.2]

15. Secondary Outcome: Overall Survival (OS) by Tumor Mutation Burden (TMB) Levels - Part 1
Description: Overall survival (OS) by tumor mutational burden (TMB) using DNA derived from tumor specimens was defined as the time from date of first treatment to the date of death due to any cause. A participant who has not died will be censored at the last known date alive.
  High TMB = ≥ 10 mutations per megabase Low TMB = < 10 mutations per megabase
Time Frame: From the date of first treatment to the date of death due to any cause (Up to approximately 72 months)
Population: All TMB evaluable participants in Part 1. Data was pre-specified to be collected only in Part 1 arm
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab+Ipilimumab
Number analyzed (Participants) | 98
Months
  High TMB (>=10 Mutations/MB): number analyzed (Participants) | 48
  High TMB (>=10 Mutations/MB) | 47.31 [14.46 to NA] — The 95% upper limit was not reached per the Kaplan-Meier method, as the probability of survival was still above 50%
  Low TMB (<10 Mutations/MB): number analyzed (Participants) | 50
  Low TMB (<10 Mutations/MB) | 11.33 [6.60 to 13.70]

16. Secondary Outcome: Progression Free Survival (PFS) by Tumor Mutation Burden (TMB) Levels - Part 1
Description: Progression Free Survival (PFS) by tumor mutational burden (TMB) using DNA derived from tumor specimens was defined as the time between the date of first dose and the first date of documented progression, as determined by blinded independent central review (BICR), or death due to any cause, whichever occurred first. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  High TMB = ≥ 10 mutations per megabase Low TMB = < 10 mutations per megabase
Time Frame: as for outcome 8
Population: All TMB evaluable participants in Part 1. Data was pre-specified to be collected only in Part 1 arm
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab+Ipilimumab
Number analyzed (Participants) | 98
Months
  High TMB (>=10 Mutations/MB): number analyzed (Participants) | 48
  High TMB (>=10 Mutations/MB) | 10.84 [3.61 to 22.21]
  Low TMB (<10 Mutations/MB): number analyzed (Participants) | 50
  Low TMB (<10 Mutations/MB) | 2.79 [1.38 to 5.39]

17. Secondary Outcome: Objective Response Rate (ORR) by Tumor Mutation Burden (TMB) Levels - Part 1
Description: Objective response rate (ORR) by tumor mutational burden (TMB) using DNA derived from tumor specimens was defined as the percentage of treated participants with confirmed complete response (CR) or partial response (PR) per RECIST 1.1 based on Blinded Independent Central Review (BICR) assessment.
  CR = Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  PR = At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  High TMB = ≥ 10 mutations per megabase Low TMB = < 10 mutations per megabase
Time Frame: From first dose up to approximately 72 months
Population: All TMB evaluable participants in Part 1. Data was pre-specified to be collected only in Part 1 arm
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab+Ipilimumab
Number analyzed (Participants) | 98
Percentage of participants
  High TMB (>=10 Mutations/MB): number analyzed (Participants) | 48
  High TMB (>=10 Mutations/MB) | 52.1 [37.2 to 66.7]
  Low TMB (<10 Mutations/MB): number analyzed (Participants) | 50
  Low TMB (<10 Mutations/MB) | 16.0 [12.1 to 34.2]

ADVERSE EVENTS:
Time Frame: Part 1: SAEs and AEs are assessed from first dose to 30 days post last dose (Up to approximately 25 months). Participants were assessed for all-cause mortality from their first dose to study completion (Up to approximately 72 months). Part 2: SAEs and AEs are assessed from first dose to 30 days post last dose (Up to approximately 25 months). Participants were assessed for all-cause mortality from their first dose to study completion (Up to approximately 59 months).
Arm/Group | Nivolumab+Ipilimumab | Nivolumab+Ipilimumab+Chemotherapy
All-Cause Mortality (participants affected / at risk) | 209/288 | 28/36
Serious Adverse Events (participants affected / at risk) | 171/288 | 26/36
Other Adverse Events (participants affected / at risk) | 282/288 | 35/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab+Ipilimumab (N=288) | Nivolumab+Ipilimumab+Chemotherapy (N=36)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 2 | 0
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac tamponade (Cardiac disorders) | 2 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 2
Myocarditis (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 3 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 2
Hyperthyroidism (Endocrine disorders) | 2 | 0
Hypophysitis (Endocrine disorders) | 3 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Autoimmune colitis (Gastrointestinal disorders) | 2 | 0
Autoimmune enteropathy (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 7 | 2
Constipation (Gastrointestinal disorders) | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 10 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1
Asthenia (General disorders) | 1 | 1
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
Gait disturbance (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 6 | 4
Sudden death (General disorders) | 2 | 1
Swelling face (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Adrenalitis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 2 | 0
Encephalitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 3 | 0
Large intestine infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 26 | 1
Sepsis (Infections and infestations) | 7 | 0
Septic shock (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Wound infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 1
Influenza B virus test positive (Investigations) | 1 | 0
Liver function test increased (Investigations) | 2 | 0
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 0
Failure to thrive (Metabolism and nutrition disorders) | 2 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 20 | 2
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain oedema (Nervous system disorders) | 1 | 0
Cerebellar infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dyskinesia (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 2
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 0
Paraneoplastic encephalomyelitis (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 2 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Mental status changes (Psychiatric disorders) | 2 | 2
Acute kidney injury (Renal and urinary disorders) | 4 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 11 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 | 0
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0
Embolism (Vascular disorders) | 3 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab+Ipilimumab (N=288) | Nivolumab+Ipilimumab+Chemotherapy (N=36)
Anaemia (Blood and lymphatic system disorders) | 67 | 12
Neutropenia (Blood and lymphatic system disorders) | 2 | 2
Adrenal insufficiency (Endocrine disorders) | 18 | 4
Hyperthyroidism (Endocrine disorders) | 25 | 4
Hypothyroidism (Endocrine disorders) | 33 | 6
Vision blurred (Eye disorders) | 17 | 2
Abdominal discomfort (Gastrointestinal disorders) | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 34 | 3
Colitis (Gastrointestinal disorders) | 10 | 3
Constipation (Gastrointestinal disorders) | 71 | 14
Diarrhoea (Gastrointestinal disorders) | 111 | 14
Dry mouth (Gastrointestinal disorders) | 32 | 2
Flatulence (Gastrointestinal disorders) | 5 | 2
Nausea (Gastrointestinal disorders) | 110 | 16
Vomiting (Gastrointestinal disorders) | 60 | 6
Asthenia (General disorders) | 17 | 0
Chills (General disorders) | 36 | 0
Fatigue (General disorders) | 159 | 20
Gait disturbance (General disorders) | 9 | 3
Influenza like illness (General disorders) | 10 | 6
Malaise (General disorders) | 6 | 4
Mucosal inflammation (General disorders) | 3 | 2
Non-cardiac chest pain (General disorders) | 19 | 0
Oedema peripheral (General disorders) | 48 | 5
Pain (General disorders) | 16 | 1
Pyrexia (General disorders) | 47 | 5
Bronchitis (Infections and infestations) | 12 | 2
Candida infection (Infections and infestations) | 6 | 2
Cellulitis (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 34 | 2
Sinusitis (Infections and infestations) | 15 | 2
Upper respiratory tract infection (Infections and infestations) | 36 | 3
Urinary tract infection (Infections and infestations) | 16 | 4
Fall (Injury, poisoning and procedural complications) | 20 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 20 | 1
Alanine aminotransferase increased (Investigations) | 27 | 3
Amylase increased (Investigations) | 34 | 4
Aspartate aminotransferase increased (Investigations) | 40 | 4
Blood alkaline phosphatase increased (Investigations) | 26 | 3
Blood creatinine increased (Investigations) | 14 | 4
International normalised ratio increased (Investigations) | 1 | 2
Lipase increased (Investigations) | 49 | 6
Lymphocyte count decreased (Investigations) | 18 | 4
Neutrophil count decreased (Investigations) | 9 | 8
Platelet count decreased (Investigations) | 5 | 5
Weight decreased (Investigations) | 66 | 7
Weight increased (Investigations) | 19 | 4
White blood cell count decreased (Investigations) | 7 | 4
Decreased appetite (Metabolism and nutrition disorders) | 95 | 9
Dehydration (Metabolism and nutrition disorders) | 24 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 26 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 19 | 4
Hypernatraemia (Metabolism and nutrition disorders) | 4 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 50 | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 19 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 41 | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 37 | 9
Hyponatraemia (Metabolism and nutrition disorders) | 62 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 16 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 84 | 13
Arthritis (Musculoskeletal and connective tissue disorders) | 8 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 57 | 6
Flank pain (Musculoskeletal and connective tissue disorders) | 9 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 17 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 25 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 | 4
Dizziness (Nervous system disorders) | 38 | 6
Dysgeusia (Nervous system disorders) | 12 | 2
Headache (Nervous system disorders) | 52 | 5
Neuropathy peripheral (Nervous system disorders) | 5 | 3
Paraesthesia (Nervous system disorders) | 15 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 12 | 3
Presyncope (Nervous system disorders) | 3 | 2
Taste disorder (Nervous system disorders) | 8 | 2
Tremor (Nervous system disorders) | 5 | 2
Anxiety (Psychiatric disorders) | 28 | 4
Confusional state (Psychiatric disorders) | 11 | 3
Depression (Psychiatric disorders) | 23 | 3
Insomnia (Psychiatric disorders) | 45 | 7
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 93 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 93 | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 16 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 22 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 35 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 19 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 17 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 24 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 17 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 41 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 88 | 17
Rash (Skin and subcutaneous tissue disorders) | 47 | 11
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 47 | 8
Hypertension (Vascular disorders) | 37 | 3
Hypotension (Vascular disorders) | 18 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/59/NCT02659059/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT02659059/SAP_001.pdf